CLINICAL TRIAL: NCT00576212
Title: The Impact of a Telephone-based Support Intervention on the Long-term Well-being of Women Undergoing Termination of Pregnancy for Fetal Anomaly
Brief Title: Impact of a Telephone-based Support Intervention on the Long-term Well-being of Women Undergoing Termination of Pregnancy for Fetal Anomaly
Acronym: TOPFA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant.
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-0157-E
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Psychological Sequelae of Termination of Pregnancy for Fetal Anomaly
Keywords: termination fetal anomaly; psychological sequelae pregnancy termination for anomalies; supportive follow-up pregnancy termination anomalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects in the intervention group will receive supportive telephone calls biweekly for 6 months.
  Interventions: Behavioral: supportive call
- B (No Intervention): Subjects in the control group will receive no intervention.

INTERVENTIONS:
Behavioral: supportive call — Each subject in the intervention group will receive a 10 minute (or longer) biweekly telephone call from a psychologist intended to provide non-judgemental support to TOPFA women with the aim of reducing depression, guilt, isolation, shame, marital discord, and other common psychological sequelae of termination for fetal anomalies.
  Arms: A

SUMMARY:
This study focuses on women undergoing termination of pregnancy for fetal anomalies (TOPFA). Psychological consequences of such terminations may be even greater than those associated with spontaneous losses of pregnancy because of shame and guilt which can result in social isolation. Currently, there is little support for women after they have left hospital. In this study, 50 TOPFA women will be randomly assigned to an intervention group and 50 to a control group. By completing four questionnaires at the time of induction of labour, total sample will be assessed for depression, stress and "hardiness"; they will be reassessed at 3, 6, and 12 months. Total sample will be interviewed by phone at 6 and 12 months. We hope to determine whether a telephone-based intervention (a biweekly supportive call) can decrease the emotional distress experienced by women undergoing termination of pregnancy.

DETAILED DESCRIPTION:
We hypothesize that: 1)women in the intervention group will show lower rates of depression and stress and a significant increase in hardiness over time at 6 and 12 months post-termination compared with the control group; 2) women who score low on hardiness initially will experience more psychological distress at 6 and 12 months than subjects who score higher initially, irrespective of group; 3) women who have anxious/avoidant attachment styles will not show an improvement in psychological distress over time, irrespective of group.

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years of age undergoing termination of pregnancy for fetal anomaly at Mount Sinai Hospital, Toronto
* fluent in oral and written English
* able to understand the nature of the study
* can provide informed consent
* can be reached by telephone

Exclusion Criteria:

-women who are currently seeing a therapist or undergoing psychiatric care, and women who do not meet all of the inclusion criteria

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
At time of induction of labour and at 3, 6, and 12 months post-TOPFA: scores on the Beck Depression Inventory, the Impact of Events Scale, the Lang and Goulet Hardiness Scale,the Relationship Scales Questionnaire | One year

SECONDARY OUTCOMES:
Total sample will be interviewed by telephone at 6 and 12 months post-TOPFA | One year

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Sloan, PhD MD FRCP, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada